CLINICAL TRIAL: NCT05970614
Title: The Effect of Eye Masks and Earplugs on Sleep Quality and Life Findings In Intensive Care Unit Patients
Brief Title: The Effect of Eye Masks and Earplugs In Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, onur çetinkaya, PhD, Lecturer, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OKU-SHMYO-OC-01
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Sleep Quality; Vital Signs
Keywords: sleep quality; vital signs; intensive care; ear plugs; eye masks
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ear Protective Devices

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with control and intervention groups
Who Masked: Participant
Masking Description: Only participants were blinded in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No application will be made to the participants. Participants will receive routine care.
- intervention group (Other): In addition to routine care, participants will be given eye masks and ear plugs for 3 days.
  Interventions: Other: Eye masks and ear plugs

INTERVENTIONS:
Other: Eye masks and ear plugs — Eye masks and ear plugs will be applied to patients for 3 days between 22:00 and 06:00.
  Arms: intervention group

SUMMARY:
This study was planned as a randomized controlled and experimental study to evaluate the effect of eye masks and earplugs on sleep quality and vital signs in intensive care patients.

DETAILED DESCRIPTION:
The research will be conducted with 60 patients hospitalized in the intensive care units of a state hospital. Research data will be collected with a questionnaire, vital signs follow-up form, insomnia severity index, and Richards-Campbell Sleep Quality Scale. Patients will be divided into intervention and control groups. Eye mask and ear plugs will be applied to the intervention group for 3 days, and the control group will receive routine care. The study will be terminated after 3 days of follow-up for each patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Able to answer all questions and communicate,
* Those who agreed to participate in the research
* Being in the category of insomnia, moderate insomnia, or severe insomnia according to the insomnia severity index,
* Not sedating
* Not connected to a ventilator
* No hearing problem
* Glasgow Coma Score of 15

Exclusion Criteria:

* Connecting to the ventilator during operation
* Sedation during the study
* Wanting to leave the research during the study
* Being in the intervention group and removing the eye patch or earplug during sleep
* GCS falling below 15

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Personal questionnaire | Only one times. At the first meeting (up to one day).
  It is a form consisting of 22 questions in order to investigate the sociodemographic characteristics and health status of the patients.
Vital signs follow-up form | up to 3 days
  It will be used to measure patients' fever, pulse, respiration, blood pressure and sPO2 values. It will be applied to patients at 22, 02, 06 hours. Also, the daily average hour will be calculated at the end of each day.
Insomnia Severity Index | up to 3 days
  It will be used to measure the severity of insomnia in patients. It consists of 7 questions and each question can receive points between 0 and 4. A maximum score of 28 and a minimum score of 0 are obtained on the scale, and as the score increases, the severity of insomnia increases.
Richards-Campbell Sleep Scale | up to 3 days
  The scale consists of 6 questions and the question is between 0 and 100 points. The higher the score, the higher the sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Osmaniye Public Hospital, Osmaniye, Merkez, Turkey (Türkiye)